CLINICAL TRIAL: NCT00055614
Title: Phase I Study of Oral Topotecan as Consolidation for Patients With Mullerian Origin Tumors (Ovary, Tube, Peritoneum)
Brief Title: Topotecan in Treating Patients With Advanced Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BIDMC-E-010405FB; CDR0000269138 (Registry Identifier: PDQ (Physician Data Query)); NEDH-E-010405FB
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2007-04

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Topotecan; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: topotecan hydrochloride
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of topotecan in treating patients who have advanced ovarian epithelial, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and duration of prolonged topotecan as maintenance in patients with advanced ovarian epithelial, fallopian tube, or primary peritoneal cancer with complete clinical response after platinum-based chemotherapy.
* Determine the safety of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral topotecan twice daily for 21 days. Treatment repeats every 28 days for up to 6 months in the absence of unacceptable toxicity or disease progression.

Patients who tolerate course 1 may receive an escalated dose of topotecan for subsequent courses. The maximum tolerated dose is defined as the dose tolerated by the majority of the patients.

Patients are followed every 2 months for at least 6 months.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal serous cancer

  * Stage IIIB, IIIC, or IV
  * Surgically staged and debulked
* Complete clinical response after first-line platinum-based chemotherapy (cisplatin or carboplatin) defined by all of the following criteria:

  * No evidence of cancer by history or physical examination
  * CA 125 no greater than 35 units/mL
  * No evidence of residual cancer on CT scan of the abdomen/pelvis and chest x-ray
* Must have received at least 5 courses of first-line chemotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count at least 1,200/mm^3
* Platelet count at least 90,000/mm^3

Hepatic

* Bilirubin normal
* ALT and AST less than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 1.5 ULN

Renal

* Creatinine clearance at least 60 mL/min

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior first-line chemotherapy
* At least 3 years since other prior chemotherapy (other than first-line chemotherapy for ovarian, fallopian tube, or primary peritoneal cancer)
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* No prior abdominopelvic radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* No concurrent surgery

Other

* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2002-05; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A. Cannistra, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States